CLINICAL TRIAL: NCT04616989
Title: Integration of Mental Health Care in Communities Affected by the COVID-19 Pandemic in Central Uganda
Brief Title: Mental Health in Communities Affected by COVID-19 in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Integration of mental health
Record Dates: First submitted 2020-10-20; First posted 2020-11-05 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Community Mental Health

STUDY DESIGN:
Intervention Model Description: Participants in the intervention arm will receive leaflets about the mental health literacy while those in the control arm will receive COVID-19 leaflets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psycho-education intervention arm (Experimental): Participants will receive psycho-education materials
  Interventions: Behavioral: Psycho-education
- Comparator arm (Active Comparator): Participants will receive COVID-19 leaflets
  Interventions: Behavioral: Comparator

INTERVENTIONS:
Behavioral: Psycho-education — Provide psycho-education to members of the community
  Arms: Psycho-education intervention arm
Behavioral: Comparator — Distribution of COVID-19 leaflets to members of the community
  Arms: Comparator arm

SUMMARY:
Introduction: During pandemics like the COVID-19, a significant number of the populace suffer from psychological distress (PD) that often abates naturally over time in the majority of people but persists in others to become pervasive and severe enough to trigger the onset of common mental disorders (CMD) like major depressive disorders (MDD), generalized anxiety disorders (GAD), post-traumatic stress disorders (PTSD) and substance misuse disorders (SUD). Once identified, psychological distress as well as CMD can be managed using psychotherapy or pharmacotherapy. However, low levels of mental health literacy (MHL) manifested by the individual's unawareness of CMD symptoms, limited human and mental health infrastructure resources and high levels of mental illness stigma (MIS), are barriers to integration of mental health care in general health care during pandemics and epidemics such as the COVID-19.

The study objectives will include: (a) Documenting MHL, PD, MDD, GAD, PTSD and SUD levels in the study population, (b) Determining the effectiveness of a psycho-education intervention delivered by village health team (VHT) members on study outcomes

Methods: We shall employ an open label cluster-randomized trial design, with each village as a cluster, to conduct the study in 24 villages (12 intervention and 12 control villages) in Kampala (n= 15), Wakiso (n= 3), Masaka (n= 2) and Mukono (n= 4) districts. To ensure balance between the two study arms, villages underwent stratified randomization on the basis of rural vs urban population. The second level of stratification will be achieved by a separate randomization procedure performed within each stratum to ensure gender balance within each cluster

We will develop information education and communication materials (IEC) aimed at improving MHL and reducing MIS. In the intervention arm (n=12 villages), VHTs will distribute the IEC materials in every 12th household till they accrue 420 individuals (adults ≥ 18 years old) who express interest in participating in the study. In the control arm (n=12 villages), VHTs will distribute MOH COVID-19 information leaflets in every 12th household till they accrue 420 individuals who express interest in participating in the study. Within 7days after distribution of the materials, trained research assistants will schedule and assess participants (through a phone interview) for MHL, PD, MDD, GAD, PTSD and SUD. Individuals who don't have phones will be asked to provide a phone number of a friend or relative through which the interviews can be conducted; interviews could also be conducted using the VHTs' phone. Cost data will be collected using available implementation data. We will document the number of individuals from both arms who will contact the investigators

Data analysis plans: We will (a) report frequencies and percentages and their 95% confidence intervals for the first objective, (b) use an intention to treat analysis to analyze the second objective,

Conclusion: Findings from this research will guide policy and practice regarding the integration of mental health services in the community in the context of epidemic preparedness and response.

DETAILED DESCRIPTION:
Study design: The investigators will use a multi-stage open-label cluster-randomized trial of 24 randomly chosen villages (n=12 intervention and n=12 control) in Kampala (n=15), Wakiso (n=3), Mukono (n=4) and Masaka (n=2) districts. Intervention and control villages are at least 20km apart to avoid contamination

Study procedure:

(i) Randomization and sampling: The investigators shall employ an open label cluster-randomized trial design, with each village as a cluster, to conduct the study in 24 villages (12 intervention and 12 control villages) in Kampala (n= 15), Wakiso (n= 3), Masaka (n= 2) and Mukono (n= 4) districts. To ensure balance between the two study arms, villages underwent stratified randomization on the basis of rural vs urban population. The second level of stratification will be achieved by a separate randomization procedure performed within each stratum to ensure gender balance within each cluster

The investigators shall employ the multistage open label sampling approach to select 840 participants from 24 randomly selected villages located in the 362 parishes (5250 villages) that span the study districts. Study villages will be selected using the probability proportional to size approach (based on number of parishes/villages per district). Thus, the investigators shall select 15 villages from Kampala district (3297 villages), 4 villages from Mukono district (813 villages), 2 villages from Masaka district (436 villages) and 3 villages from Wakiso district (704 villages). The villages are at least 20km apart to avoid contamination (individuals interacting during the intervention).

(ii) Participant identification: The investigators shall engage the VHT and village Local Chairpersons to distribute leaflets describing the study to every 12th household in their catchment area till they accrue 38 participants in their village who express interest in participating in the study. This figure is based on an average of 4710 households per village. Thus 4710/38 is approximately every 12th household. Individuals who express interest in the study will be given 2 consent forms which they will read and sign should they decide to participate; they will retain one copy. VHTs will read out the consent form to individuals who can neither read nor write and obtain informed consent (participants will use their thumb print soaked in an inkpad to consent). Consent forms will be translated into Luganda. The VHT will then get the participant's telephone contact and provide it to the project administrator who will pass them to research assistants. Individuals who don't have phones will be asked to provide a phone number of a friend or relative through which the interviews can be conducted- interviews could also be conducted using the VHTs' phone if the participants comfortable receiving calls on the VHT's telephone. The VHT will inform the project administrator of participants without personal phones and indicate how that participant can be contacted. The investigators will conduct a times and motions assessment to document the duration of the interventions as well as the amount of money spent on transport refunds for the VHTs and the airtime costs

(iii) Baseline data collection: Trained research assistants will call participants and schedule a phone interview and collect demographic (age, gender, education level and place of residence) information and administer the Mental health Knowledge Schedule (MAKS) to assess for MHL, Kesler-10 (K-10) to measure PD, the Generalized Anxiety Disorder scale (GAD-7) to assess for GAD, Patient Health Questionnaire-9 (PHQ-9) to assess for MDD Post-Traumatic Stress Disorder- Primary Care Screen (PTSD-PC) for PTSD and the Alcohol Smoking and Substance Involvement screening Test (ASSIST) to assess for SUD.

(iv) The intervention: Within a week of the baseline surveys, VHTs in the 12 intervention villages described above- (a) basic information about the symptoms of PD (b) their adverse effects, (c) the signs and symptoms of CMD, (d) the benefits associated with having them treated and (e) the contact details of the research team should they need more information. See a template of the IEC materials attached. Previous studies have administered the post-test questionnaires a week after the baseline assessment .

In the 12 control villages, VHTs will distribute the MOH IEC materials that contain information about (a) the signs and symptoms of the COVID-19 and the preventive measures, (b) the fact that individuals may suffer from PD during the pandemic (c) the sources from where they can get psychosocial help and (d) the contact details of the research team should they need more information. The IEC materials will be distributed to individuals who participated in the baseline surveys

Mitigating the possibility of contamination between the study arms: Being an educational intervention, there is a chance that participants in the control villages will access IEC materials distributed to those in the intervention arm, leading to contamination of the study findings. To avoid contamination, the investigators will do the following: (i) randomize villages so that they are at least 20km apart (with the limited human movements during the COVID-19 pandemic, we anticipate that there will be little by way of people sharing the IEC materials), (ii) conduct the assessments within a week of distributing the materials to limit the chances that the information will be widely circulated, (iii) ask participants in the control arms if they accessed the IEC materials meant for the control group.

(v) Follow-up data collection: Within a week after the VHTs have distributed IEC materials, research assistants will call participants from both arms and (i) confirm whether they received IEC materials (and read it), then (ii) schedule a phone interview to administer the instruments administered at baseline (MAKS, K-10, GAD-7, PHQ-9, PTSD-PC and ASSIST).

Study measures: Research assistants will administer standardized questionnaires to collect: i) Demographic variables including age, gender, physical address, contact information, marital and employment status, education level ii) primary study variable (MHL using MAKS) and (iii) secondary variables including PD using the K-10, GAD using the GAD-7, MDD using the PHQ-9, PTSD using the PTSD-PC and SUD using the ASSIST.

Participant Follow-up: Participants will be assessed for the outcomes of interest at baseline and within a week (7 days). Participants who have been referred to the psychosocial teams will be called after 14 days to find out whether they followed up on the referral and if not, state the reasons for not doing so.

Adverse event reporting during the interviews: The investigators anticipate that there will be minimal adverse events that are directly related to the study, mainly psychological distress resulting from answering the questions during the survey or loss of private data. However, in the event that the investigators realize any severe form of distress, or loss of privacy/confidentiality, then the investigators will report it promptly reported to the SOMREC/UNCST.

Community tracing: In the event that a participant cannot be accessed for the second interview after the baseline one, then, the investigators will ask the VHT to visit the physical location and find out the reason for non-response. The VHT will be provided with a Log to record this kind of information which could be loss of a phone, change in phone number of withdrawal from the study among other reasons. If the participant can't be contacted on phone and physically, (may have moved house), then the investigators will consider this a loss to follow up.

Sample size and statistical considerations Hypothesis: The investigators hypothesize that (a) the MHL levels are low in the communities in comparison to those observed in high income countries, (b) a psycho-education intervention delivered by VHTs will lead to a 50% increase in MHL levels in the intervention arm compared to the control arm (that this difference will be clinically significant), (c) more participants in the intervention arm will contact the study team compared to the control arm - and that this difference will be clinically significant

1. Sample size for objective 1. To document the baseline community MHL level, the investigators will use the Leslie-Kish formular for calculating the sample size for cross sectional studies. The formula states that: n = Z2 p (1-p)/E2. n- sample size, E-The standard error (5%), p- Proportion of patients; 50%.The prevalence was estimated at 50% as the conservative estimates for outcomes or effects sizes with limited literature to refer to (in this case, prevalence of poor MHL in the Ugandan community). Z- The standard normal deviation of 1.96 corresponding to 95% confidence interval Substituting; n=1.962 X 0.5 X (1-0.5)/0.052 n= 384. b) For the population survey, the investigators will use the sample size calculation, but use a community correction effect of 2. Thus the sample size for the community sample will be 384X2 = 764. The investigators will add a 10% sample size to cater for incomplete data mainly due to failure to complete an interview. Thus, the total sample size will be 840 participants (420 in the control and 420 in the intervention arms).
2. Sample size for objective 2: To determine the effectiveness of the psycho-education intervention, the investigators have calculated the size of effects that the sample will be able to detect a clinically significant difference in MHL level between the intervention and control arms. The nature of the educational intervention makes randomization by clusters (villages) more appropriate in comparison to randomization by individuals or household.

To estimate the number of villages required per arm for a clinically significant effect size of 50%: The investigators assume power of 80% at the 95% confidence level, mean MHL score of 14.14 and standard deviation (SD) of 2.19, cluster-size of 35 participants and coefficient of variation of 0.25, which yields ~8 villages per trial-arm. The investigators shall include a minimum of 12 villages per arm (50% increment) to cater for the following limitations; i) the large proportion of participants who do not own mobile phones (~30%) (Incomplete data due to participants not being able to complete interviews). Therefore, 24 villages (both arms) will be required; thus, including up to 840 participants (420 per trial-arm).

Data collection and management: Data will be collected on paper and then entered into a centralized, web-based data management scheme using the open source software REDCap™.

Statistical Analysis

Objective 1: The investigators will report frequencies and percentages of the study outcomes and their 95% confidence intervals.

Objective 2: An intention-to-treat analysis will be conducted to compare the groups at baseline and within 4 weeks to assess the effects of the intervention on MHL. The dependent variable (MHL) will be calculated as a continuous variable. Independent variables including presence of PD, MDD, GAD, PTSD or SUD will be presented as continuous and categorical variables. Baseline characteristics of the intervention and control arms will be compared at the 5% level to assess if successful randomization was achieved. Data on potential confounders and effect modifiers, including variables that fail to achieve successful randomization (e.g. socio-demographic parameters) shall be used to control for confounding and effect modification. Between-subject analysis at week 4 will be used to assess the direct effect of the intervention by determining if there is a significant difference between the mean MHL scores in the intervention and control arms. Within-subject analysis will be performed among patients in the intervention arm by applying the Generalized Estimating Equations method on repeated measures data.

Data safety management board: The data safety management board (DSMB) will be comprised of Prof Eugene Kinyanda (Psychiatrist and Senior Epidemiologist), Dr Moses Ocan (pharmacologist and IRB member), and Dr. Paul Bangirana (Clinical psychologist with vast experience in conducting RCT) from Makerere University. The PI will have periodic meetings with the DSMB and provide them with reports about the study activities using an agreed template. There will be at least two meetings during the study period one at the beginning and another midway through the study. Members of the DSMB will make a visit at the Butabika Hospital where data will be collected (phone calls) and stored. During this visit, the study procedures (SOPs and manuals), study responsibilities (delegation log), site facilities (call rooms/data room), study materials (stationary and administrative materials) and the recruitment and retention plan will be discussed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and above who live in the community where data will be collected

Exclusion Criteria:

* Individuals with acute illnesses that will prevent them from providing information during data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 814 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Change in mental health literacy | 2 months
  We will document the change in the mean scores of mental health literacy between the two arms measured using the Mental health Knowledge Schedule (MAKS) instrument

SECONDARY OUTCOMES:
Burden of anxiety disorders in the community | 2 months
  We will document the prevalence of anxiety using the GAD instrument in the 2 arms
Burden of PTSD in the community | 2 months
  We will document the prevalence of PTSD using the PTSD-PC instrument in the 2 arms
Burden of substance use disorders in the community | 2 months
  We will document the prevalence of substance use disorders using the ASSIST instrument in the 2 arms
Burden of depression disorders in the community | 2 months
  We will document the prevalence of depression use disorders using the PHQ-9 instrument in the 2 arms

CONTACTS AND LOCATIONS:
Locations (1):
- Dickens Akena, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akena D, Kiguba R, Muhwezi WW, Kwesiga B, Kigozi G, Nakasujja N, Lukwata H. The effectiveness of a psycho-education intervention on mental health literacy in communities affected by the COVID-19 pandemic-a cluster randomized trial of 24 villages in central Uganda-a research protocol. Trials. 2021 Jul 13;22(1):446. doi: 10.1186/s13063-021-05391-6. PMID 34256810